CLINICAL TRIAL: NCT02965274
Title: An Open Label, Randomized, 2-Period, 2-Treatment,2-Sequence, Crossover, Single-Dose BE of Fluoxetine Tablets 20 mg [Torrent,India] Versus Sarafem 20 mg Tablet [ Warner Chilcott LLC, USA] in Healthy Subjects-Fed Condition.
Brief Title: Bioequivalence Study of Torrent Pharmaceuticals Ltd.'s Fluoxetine Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK-12-057
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Torrent's Fluoxetine Tablets 20 mg
  Interventions: Drug: Torrent's Fluoxetine Tablets
- Reference (Active Comparator): Warner Chilcott LLC, USA
  Interventions: Drug: Warner Chilcott LLC's Sarafem Tablet

INTERVENTIONS:
Drug: Torrent's Fluoxetine Tablets
  Arms: Test
Drug: Warner Chilcott LLC's Sarafem Tablet
  Arms: Reference

SUMMARY:
Subjects to compare the single dose bioavailability of Torrent's Fluoxetine Tablets 20 mg and Sarafem® 20 mg Tablets of Warner Chilcott LLC, USA. Dosing periods of studies were separated by a washout period of 35 days.

DETAILED DESCRIPTION:
An Open Label, Randomized, 2-period, 2- Treatment, 2-Sequence, Crossover, Single-dose Bioequivalence Study of Fluoxetine Tablets containing Fluoxetine 20 mg ( Test Formulation, Torrent Pharmaceutical Ltd., India) Versus Sarafem® 20 mg Tablets containing Fluoxetine 20 mg (Reference, Warner Chilcott LLC, USA) in Healthy Human Volunteers Under Fed Condition.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male
* Age: 18-45 years (inclusive both)
* Volunteer with BMI of 18.5-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day.

Exclusion Criteria:

* Inability to communicate or co-operate.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of pre-existing bleeding disorder.
* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* HIV, HCV, HBsAg positive volunteers.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* Participation in any study within past 3 months,
* History of alcohol or drug abuse.
* History of consumption of prescribed medication since last 14days or OTC medication/ herbal remedies since last 7 days before beginning of the study. Positive to Breath alcohol test.
* Positive to breath alcohol test.
* Volunteer found to be positive for Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, Cocaine positive volunteers based on urine test.
* Systolic blood pressure less than 100 mmHg or more than 139 mmHg and diastolic blood pressure less than 60 mm Hg or more than 89 mm Hg.
* Pulse rate less than 60/minute or more than 100/minute.
* Oral temperature less than 95°F or more than 98.9°F.
* Respiratory rate less than 10/minute or more than 20/minute.
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* Recent History of kidney or liver dysfunction.
* Volunteers suffering from any psychiatric (acute or chronic) disorder.
* Existence of any surgical or medical condition, which, in the judgment of the Chief Investigator and/or clinical investigator/physician, might interfere with the absorption; distribution,· metabolism or excretion of the drug or likely to compromise the safety of Volunteers.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose to 72 hours post-dose
AUC | pre-dose to 72 hours post-dose

IPD SHARING:
Plan to Share IPD: No